CLINICAL TRIAL: NCT04389021
Title: Clinical Effectiveness of Virtual Reality Simulation in Reducing Discomfort, Anxiety and Pain During Intrauterine Device Insertion: A Randomized Clinical Trial
Brief Title: Virtual Reality Simulation for Intrauterine Device Insertion: A Randomized Clinical Trial
Acronym: VR-IUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Dirk Timmerman, Clinical Head Gynecology, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: S63124
Record Dates: First submitted 2020-05-06; First posted 2020-05-15 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2020-05

CONDITIONS: IUD
Keywords: Virtual Reality; IUD; Discomfort

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR (Experimental): The intervention group will receive VR support upon the standard of care during the procedure.
  Interventions: Device: Virtual Reality
- Control (No Intervention): The control group will have standard care without the VR support.

INTERVENTIONS:
Device: Virtual Reality — The VR goggles have a 2560×1440 5.5" (538ppi) fast-switching LCD screen with standard 60Hz refresh, "overclocked" 72Hz refresh, running Android 7.1.2 Nougat with a Quad-core Qualcomm Snapdragon 821 (two 2.3GHz Kryo HP cores and two 2.15GHz Kryo cores). Adreno 530 as GPU. It is 190 x 105 x 115 mm en weighs 470 g (1.04 lbs). The goggles have built-in speakers, a controller, proximity sensor, 3DOF sensors (both headset and controller).
  Any pre-procedural self-administration of pain medication will be recorded. Trained staff-members or senior residents will do all IUD insertions, according to the local protocol.
  Arms: VR

SUMMARY:
Aim of this study is to evaluate the effect of VR on the patients overall experience during the IUD insertion procedure.

DETAILED DESCRIPTION:
A single center, investigator initiated randomized controlled clinical trial. 200 women to be recruited, 100 in the intervention group and 100 in the control group.

The control group will receive the usual treatment (without specific pain management) and the intervention group will receive the usual treatment with VR support.

Endpoints are:

* Objective: successful procedure, need for general anesthesia, presence of syncope and/or vomitus
* Subjective: Pain, procedural cooperation, the degree of difficulty encountered by the physician in performing the treatment, ability to complete VR procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women who are seeking hormonal intrauterine contraception will be offered participation in the trial if they are 18 years of age or older (minors can be included if a guardians permission has been obtained), are not pregnant, and are willing to follow-up after 6 weeks for a sonographic IUD check.

Exclusion Criteria:

* Epilepsy
* Auditive or visual disabilities
* Invalidating claustrophobia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Patients overall experience of IUD insertion | At insertion
  Primary outcome of this study is the patients overall experience of the insertion / replacement of a hormonal IUD. This will be measured by using a Visual Analog Scale (0-100mm, continuous scale). The left extreme of this scale represents no distress, and the right extreme represents unbearable distress.

SECONDARY OUTCOMES:
Pain during insertion | At insertion and 6 weeks later
  Assessment of the effect of VR support on pain by the Numeric Pain Rating Scale (0-100), the higher the score, the more pain.
Discomfort | At insertion and 6 weeks later
  Assessment of the degree of discomfort of the treatment procedure by the patient, by mean of a Visual analogue scale (0-100mm, continuous scale).
Degree of difficulty encountered by the physician | At insertion
  Assessment of the degree of difficulty encountered by the physician in performing the treatment, by means of a 5-point Likert scale (1=very easy, 2=easy, 3=neutral, 4=difficult, 5=very difficult).
Success rate of the procedure | At insertion and 6 weeks later
  Assessment of the success of the procedure, by recording the correct/ incorrect position of the IUD (including expulsions and perforations) and possible need to repeat the procedure under general anesthesia. Correct placement is defined as the presence of the IUD completely within the uterine cavity visualized by ultrasound.
Patient satisfaction on the longer term | 6 weeks after insertion
  Assessment of the patient satisfaction on the longer term by asking the patient whether knowing now about the discomfort, they would repeat the procedure or recommend it to a friend. This will be assessed by using a 5-point Likert scale (1=Definitely, 2= might, 3= uncertain, 4= probably not, 5= definitely not).
Side events | At insertion
  Record of the known side events of this intervention (syncope, vomitus).

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No